CLINICAL TRIAL: NCT03462056
Title: Pilot Study of Ready to Use Therapeutic Food to Promote Weight Gain in Cystic Fibrosis
Brief Title: Ready to Use Therapeutic Food (RUTF) to Promote Growth in Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201712139
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CF Ready to Use Supplemental Food. (Experimental): Participants will receive Cystic Fibrosis Ready to Use Supplemental Food sufficient to provide approximately 20% of estimated daily caloric needs up to 500kcal of total calories, 18.5 grams of protein and 28g of fat. The supplement is also optimized to provide excellent protein quality and optimal polyunsaturated fatty acid composition
  Interventions: Dietary Supplement: Cystic Fibrosis Ready to Use Supplemental Food

INTERVENTIONS:
Dietary Supplement: Cystic Fibrosis Ready to Use Supplemental Food — Specially formulated for use by children with Cystic Fibrosis

SUMMARY:
Children with cystic fibrosis require increased caloric intake to maintain appropriate growth, an important determinant of long-term outcomes. This study seeks to determine the feasibility of using a novel therapeutic food to promote weight gain and growth in children with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis diagnosed by sweat test or genetic testing.
* Exocrine Pancreatic Insufficiency and receiving pancreatic enzyme replacement therapy
* BMI or weight for age of less than the 50th percentile

Exclusion Criteria:

* Cystic fibrosis related diabetes mellitus
* Cystic fibrosis related liver disease.
* Anaphylactic or other allergy to peanut, cow's milk, oat flour or other RUTF ingredients.
* Patients who are status-post lung or liver transplantation
* Currently receiving enteral supplemental nutrition through gastrostomy or nasogastric tube.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
BMI Z-score | 3 months
  Change in BMI Z-score

SECONDARY OUTCOMES:
Weight Z-score | 3 months
  Change in Weight Z-score
Body Composition | 3 months
  Percent body fat mass and lean mass as measured by air displacement plethysmography
Body Composition | 3 months
  Percent body fat mass and lean mass as estimated by skinfold measurements (triceps and subscapular)
Pulmonary Function | 3 months
  Change in percent estimated forced expiratory volume at one second (FEV1), and forced vital capacity (FVC)
Compliance of taking supplemental food | 3 months
  Percent consumed as compared to amount recommended.
Quality of Life | 3 months
  Cystic Fibrosis Questionnaire-Revised (CFQ-R)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan T Pitman, M.D., Principal Investigator — Washington University School of Medicine; Mark J Manary, M.D., Study Chair — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States